CLINICAL TRIAL: NCT03852017
Title: IMMERSE PC: Investigating Mindfulness and Music to Ease Radiation Side Effects in Prostate Cancer
Brief Title: Investigating Mindfulness and Music to Ease Radiation Side Effects in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Victorson, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00200537
Record Dates: First submitted 2018-12-12; First posted 2019-02-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; mindfulness; music
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Following implementation pre-testing, we will use a pilot randomized-controlled design to compare 2 groups: Group A: Mindfulness (n=25), a daily audio-session, which teaches emotional self-regulation skills through the adoption of mindful awareness practices into one's life; and Group B: Relaxing Music (n=25) - a daily audio session of peaceful and relaxing music. Participants will be assessed at baseline just prior to randomization to the two study arms (T1), followed by assessments at the end of the intervention period (T2), and 1 month (T3) and 3 months (T4) after the 4-week intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Audio Program (Experimental): Mindfulness Audio Program is a daily audio-session, which teaches emotional self-regulation skills through the adoption of mindful awareness practices into one's life
  Interventions: Behavioral: Audio Program
- Music Audio Program (Active Comparator): Music Audio Program is a daily audio session of peaceful and relaxing music
  Interventions: Behavioral: Audio Program

INTERVENTIONS:
Behavioral: Audio Program

SUMMARY:
In this study, the researchers will examine the implementation feasibility, acceptability, and initial effects of a brief eHealth mindfulness intervention, compared to brief relaxing music, to reduce self-reported symptoms of fatigue, anxiety, depression and sleep disturbance in a sample of localized prostate cancer patients during the receipt of radiation therapy.

DETAILED DESCRIPTION:
Eligible patients will be recruited from Northwestern Medicine's Department of Radiation Oncology and Northwestern Memorial Hospital. Participants will complete an online questionnaire prior to beginning the intervention. Following implementation pre-testing, the intervention will begin on Week 2 of radiation therapy and last 4 weeks. Upon arrival for their treatment visit, they will receive the audio program from the clinic staff. They will start the program prior to their treatment. Participants will be asked to listen to the audio-program during their radiation treatment visits, using a Bluetooth-enabled MP3 player with speaker instead of headphones or earbuds because they are not permitted during radiation therapy. The patient's ears need to be free to hear a possible communication from the radiation therapists if need be. Audio program recordings will run 3-12 minutes. Participants will turn off the program after their audio session has ended and return the audio program to the clinic staff after their treatment visit. Participants will complete an online question immediately after completing the intervention, and again 1 and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically localized prostate cancer
* Will receive at least 7 weeks of daily radiation therapy
* At least 18 years of age
* Able to speak and understand English
* Cognitively intact and free of serious psychiatric illness (as determined by referring physician)

Exclusion Criteria:

- Regular user of mindfulness meditation, which is defined as ≥ 3 times a week for the past 4 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Implementation feasibility measured by enrollment rate | Baseline
  This indicator of implementation feasibility for the program being delivered is defined by the overall enrollment rate being >/= 70% (e.g., total number of individuals enrolled/total number approached).
Implementation feasibility measured by retention rate | Throughout study completion, a total of four months.
  This indicator of implementation feasibility for the program delivered is defined by the retention rate being >/=70% (e.g., total number of individuals who remained in the trial until the end of requested participation/total number of individuals enrolled).
Implementation feasibility measured by intervention adherence | Throughout the study intervention period, a total of 4 weeks.
  This indicator of implementation feasibility for the program delivered is defined by an adherence rate of >/=70% of all possible listening opportunities during the study intervention period.
Program acceptability measured by a post-program survey at 4-weeks | Week 4
  Program acceptability will be assessed using a brief, Likert-type survey assessing participant enjoyment, satisfaction, perceived benefit, and ease of use. Acceptability is defined as ≥70% of survey responses in affirmation of this.

SECONDARY OUTCOMES:
Significant change in fatigue using the PROMIS Fatigue questionnaire | baseline; Week 4; Month 1; Month 3
  Participants were administered the PROMIS Fatigue questionnaire. Significant change was indicated by a p<.05 on fatigue scores between baseline and follow up time points between study arms.
Significant change in anxiety using the PROMIS Anxiety questionnaire | baseline; Week 4; Month 1; Month 3
  Participants were administered the PROMIS Anxiety questionnaire. Significant change was indicated by a p<.05 on anxiety scores between baseline and follow up time points between study arms.
Change in depression using the PROMIS Depression questionnaire | baseline; Week 4; Month 1; Month 3
  Participants were administered the PROMIS Depression questionnaire. Significant change was indicated by a p<.05 on depression scores between baseline and follow up time points between study arms.
Change in sleep using the PROMIS Sleep Disturbance questionnaire | baseline; Week 4; Month 1; Month 3
  Participants were administered the PROMIS Sleep Disturbance questionnaire. Significant change was indicated by a p<.05 on sleep disturbance scores between baseline and follow up time points between study arms.
Change in uncertainty intolerance using the Intolerance for Uncertainty Scale | baseline; Week 4; Month 1; Month 3
  Participants were administered the Intolerance for Uncertainty questionnaire. Significant change was indicated by a p<.05 on uncertainty intolerance scores between baseline and follow up time points between study arms.
Change in fear of recurrence using the MAX-PC Fear of Recurrence sub-scale | baseline; Week 4; Month 1; Month 3
  Participants were administered the MAX-PC Fear of Recurrence questionnaire. Significant change was indicated by a p<.05 on fear of recurrence scores between baseline and follow up time points between study arms.
Change in mindfulness using the Mindful Attention Awareness Scale | baseline; Week 4; Month 1; Month 3
  Participants were administered the Mindful Attention Awareness Scale. Significant change was indicated by a p<.05 on mindfulness scores between baseline and follow up time points between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, PhD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkey FJ. Managing the adverse effects of radiation therapy. Am Fam Physician. 2010 Aug 15;82(4):381-8, 394. PMID 20704169
- [Background] Jereczek-Fossa BA, Santoro L, Alterio D, Franchi B, Fiore MR, Fossati P, Kowalczyk A, Canino P, Ansarin M, Orecchia R. Fatigue during head-and-neck radiotherapy: prospective study on 117 consecutive patients. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):403-15. doi: 10.1016/j.ijrobp.2007.01.024. Epub 2007 Mar 29. PMID 17398020
- [Background] Jereczek-Fossa BA, Marsiglia HR, Orecchia R. Radiotherapy-related fatigue. Crit Rev Oncol Hematol. 2002 Mar;41(3):317-25. doi: 10.1016/s1040-8428(01)00143-3. PMID 11880207
- [Background] Groenvold M, Petersen MA, Idler E, Bjorner JB, Fayers PM, Mouridsen HT. Psychological distress and fatigue predicted recurrence and survival in primary breast cancer patients. Breast Cancer Res Treat. 2007 Oct;105(2):209-19. doi: 10.1007/s10549-006-9447-x. Epub 2007 Jan 3. PMID 17203386
- [Background] Kawase E, Karasawa K, Shimotsu S, Izawa H, Hirowatari H, Saito AI, Ito K, Horikawa N. Estimation of anxiety and depression in patients with early stage breast cancer before and after radiation therapy. Breast Cancer. 2012 Apr;19(2):147-52. doi: 10.1007/s12282-010-0220-y. Epub 2010 Sep 3. PMID 20814770
- [Background] Society AC. American Cancer Society Cancer Facts & Figures. Atlanta: American Cancer Society; 2014
- [Background] Garrett K, Dhruva A, Koetters T, West C, Paul SM, Dunn LB, Aouizerat BE, Cooper BA, Dodd M, Lee K, Wara W, Swift P, Miaskowski C. Differences in sleep disturbance and fatigue between patients with breast and prostate cancer at the initiation of radiation therapy. J Pain Symptom Manage. 2011 Aug;42(2):239-50. doi: 10.1016/j.jpainsymman.2010.11.010. Epub 2011 Mar 31. PMID 21454042
- [Background] Knapp K, Cooper B, Koetters T, Cataldo J, Dhruva A, Paul SM, West C, Aouizerat BE, Miaskowski C. Trajectories and predictors of symptom occurrence, severity, and distress in prostate cancer patients undergoing radiation therapy. J Pain Symptom Manage. 2012 Oct;44(4):486-507. doi: 10.1016/j.jpainsymman.2011.10.020. Epub 2012 Jul 7. PMID 22771128
- [Background] Miaskowski C, Paul SM, Cooper BA, Lee K, Dodd M, West C, Aouizerat BE, Dunn L, Swift PS, Wara W. Predictors of the trajectories of self-reported sleep disturbance in men with prostate cancer during and following radiation therapy. Sleep. 2011 Feb 1;34(2):171-9. doi: 10.1093/sleep/34.2.171. PMID 21286498
- [Background] Mohamed NE, Bovbjerg DH, Montgomery GH, Hall SJ, Diefenbach MA. Pretreatment depressive symptoms and treatment modality predict post-treatment disease-specific quality of life among patients with localized prostate cancer. Urol Oncol. 2012 Nov-Dec;30(6):804-12. doi: 10.1016/j.urolonc.2011.02.002. Epub 2011 Jul 27. PMID 21795078
- [Background] Monga U, Garber SL, Thornby J, Vallbona C, Kerrigan AJ, Monga TN, Zimmermann KP. Exercise prevents fatigue and improves quality of life in prostate cancer patients undergoing radiotherapy. Arch Phys Med Rehabil. 2007 Nov;88(11):1416-22. doi: 10.1016/j.apmr.2007.08.110. PMID 17964881
- [Background] Vadiraja HS, Rao MR, Nagarathna R, Nagendra HR, Rekha M, Vanitha N, Gopinath KS, Srinath BS, Vishweshwara MS, Madhavi YS, Ajaikumar BS, Bilimagga SR, Rao N. Effects of yoga program on quality of life and affect in early breast cancer patients undergoing adjuvant radiotherapy: a randomized controlled trial. Complement Ther Med. 2009 Oct-Dec;17(5-6):274-80. doi: 10.1016/j.ctim.2009.06.004. Epub 2009 Oct 28. PMID 19942107
- [Background] Portenoy RK. Cancer-related fatigue: An immense problem. Oncologist. 2000;5(5):350-2. doi: 10.1634/theoncologist.5-5-350. No abstract available. PMID 11040269
- [Background] Portenoy RK, Itri LM. Cancer-related fatigue: guidelines for evaluation and management. Oncologist. 1999;4(1):1-10. PMID 10337366
- [Background] Kim YH, Kim HJ, Ahn SD, Seo YJ, Kim SH. Effects of meditation on anxiety, depression, fatigue, and quality of life of women undergoing radiation therapy for breast cancer. Complement Ther Med. 2013 Aug;21(4):379-87. doi: 10.1016/j.ctim.2013.06.005. Epub 2013 Jul 6. PMID 23876569
- [Background] Lengacher CA, Johnson-Mallard V, Barta M, Fitzgerald S, Moscoso MS, Post-White J, Jacobsen PB, Molinari Shelton M, Le N, Budhrani P, Goodman M, Kip KE. Feasibility of a mindfulness-based stress reduction program for early-stage breast cancer survivors. J Holist Nurs. 2011 Jun;29(2):107-17. doi: 10.1177/0898010110385938. Epub 2010 Nov 1. PMID 21041554
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Gross CR, Kreitzer MJ, Reilly-Spong M, Wall M, Winbush NY, Patterson R, Mahowald M, Cramer-Bornemann M. Mindfulness-based stress reduction versus pharmacotherapy for chronic primary insomnia: a randomized controlled clinical trial. Explore (NY). 2011 Mar-Apr;7(2):76-87. doi: 10.1016/j.explore.2010.12.003. PMID 21397868
- [Background] Bishop SR, Lau M, Shapiro S, et al. Mindfulness: A Proposed Ooperational Definition. Clinical Psychology: Science and Practice. 2004 2004;11(3):230-241
- [Background] Hulsheger UR, Alberts HJ, Feinholdt A, Lang JW. Benefits of mindfulness at work: the role of mindfulness in emotion regulation, emotional exhaustion, and job satisfaction. J Appl Psychol. 2013 Mar;98(2):310-25. doi: 10.1037/a0031313. Epub 2012 Dec 31. PMID 23276118
- [Background] Kabat-Zinn J. Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. New York: Dell Publishing; 1990
- [Background] Victorson D, Du H, Hankin V, et al. MINDFULNESS BASED STRESS REDUCTION DECREASES FEAR OF PROGRESSION OVER TIME FOR MEN WITH PROSTATE CANCER ON ACTIVE SURVEILLANCE: RESULTS FROM A RANDOMIZED CLINICAL TRIAL. The Journal of Urology. 2012 2012;187(4S):384
- [Background] Victorson DK, M.; Maletich, C.; Lawton, R.C.; Hankin Kaufman, V.; Borrero, M.; Languido, L.; Lewett, K.; Pancoe, H.; Berkowitz, C. . A Systematic Review and Meta-Analysis of Mindfulness-Based Randomized Controlled Trials Relevant to Lifestyle Medicine. . American Journal of Lifestyle Medicine. 2014
- [Background] Vago DR, Silbersweig DA. Self-awareness, self-regulation, and self-transcendence (S-ART): a framework for understanding the neurobiological mechanisms of mindfulness. Front Hum Neurosci. 2012 Oct 25;6:296. doi: 10.3389/fnhum.2012.00296. eCollection 2012. PMID 23112770
- [Background] Moore A, Gruber T, Derose J, Malinowski P. Regular, brief mindfulness meditation practice improves electrophysiological markers of attentional control. Front Hum Neurosci. 2012 Feb 10;6:18. doi: 10.3389/fnhum.2012.00018. eCollection 2012. PMID 22363278
- [Background] Jha AP, Krompinger J, Baime MJ. Mindfulness training modifies subsystems of attention. Cogn Affect Behav Neurosci. 2007 Jun;7(2):109-19. doi: 10.3758/cabn.7.2.109. PMID 17672382
- [Background] Tang YY, Ma Y, Wang J, Fan Y, Feng S, Lu Q, Yu Q, Sui D, Rothbart MK, Fan M, Posner MI. Short-term meditation training improves attention and self-regulation. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17152-6. doi: 10.1073/pnas.0707678104. Epub 2007 Oct 11. PMID 17940025
- [Background] Larson MJ, Steffen PR, Primosch M. The impact of a brief mindfulness meditation intervention on cognitive control and error-related performance monitoring. Front Hum Neurosci. 2013 Jul 9;7:308. doi: 10.3389/fnhum.2013.00308. eCollection 2013. PMID 23847491
- [Background] Dumville JC, Hahn S, Miles JN, Torgerson DJ. The use of unequal randomisation ratios in clinical trials: a review. Contemp Clin Trials. 2006 Feb;27(1):1-12. doi: 10.1016/j.cct.2005.08.003. Epub 2005 Oct 19. PMID 16236557
- [Background] Wyatt G, Sikorskii A, Rahbar MH, Victorson D, Adams L. Intervention fidelity: aspects of complementary and alternative medicine research. Cancer Nurs. 2010 Sep-Oct;33(5):331-42. doi: 10.1097/NCC.0b013e3181d0b4b7. PMID 20467309
- [Background] Lai J-S, Cella D, Choi S, Teresi JA, Hays RD, Stone AA. Developing a fatigue item bank for the Patient-Reported Outcomes Measurement Information System (PROMIS FIB version 1). Presented at the Meeting of the Survey Methods in Multicultural, Multinational, and Multiregional Contexts (3MC), Berlin, Germany. 2008
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Flynn KE, Shelby RA, Mitchell SA, Fawzy MR, Hardy NC, Husain AM, Keefe FJ, Krystal AD, Porter LS, Reeve BB, Weinfurt KP. Sleep-wake functioning along the cancer continuum: focus group results from the Patient-Reported Outcomes Measurement Information System (PROMIS((R))). Psychooncology. 2010 Oct;19(10):1086-93. doi: 10.1002/pon.1664. PMID 20013938